CLINICAL TRIAL: NCT01762215
Title: Policy on Optimized Epilepsy Management: The Use of an Online Social Media Platform to Collect Patient-Entered Data in the Veteran Population
Brief Title: Policy on Optimal Epilepsy Management
Acronym: POEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern California Institute of Research and Education (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Veterans Administration Epilepsy Centers of Excellence (ECoE) (U.S. Federal Agency); University of California, San Francisco (Other); PatientsLikeMe (Other); UCB Pharma (Industry)
Responsible Party: Principal Investigator, Dr. John Hixson, Assistant Professor of Clinical Neurology, San Francisco Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: POEM
Record Dates: First submitted 2012-12-28; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Epilepsy; Seizure Disorder
Keywords: Epilepsy; Seizure; Veteran
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLM (Experimental): Upon consenting to the study, participants will be asked to register an account on PatientsLikeMe; no personal identifiers will be required. As part of registration patients create a user name and password for the website and share their email with PatientsLikeMe. Participants will be asked to provide a set of demographic variables and to complete a survey assessing elements of self-management, disease knowledge, social support, and quality of life. Paticipants will then use the PatientsLikeMe website for 6 weeks as much as they wish. After 6 weeks the participants are asked to complete a second survey.
  Interventions: Behavioral: PatientsLikeMe.com

INTERVENTIONS:
Behavioral: PatientsLikeMe.com — PatientsLikeMe (PLM, www.patientslikeme.com) is an established medical social networking website that encourages patients with chronic medical conditions to voluntarily share their story and seek support from a common community. Additionally, PatientsLikeMe is actively exploring opportunities to allow patients to report and track important medical data points with the hope that this will improve their longitudinal care. PatientsLikeMe has developed custom functionality for the epilepsy population including seizure tracking, peer support, and printable doctor visit support sheets.
  Other Names: PLM; www.patientslikeme.com

SUMMARY:
This study examines the use of an online social media platform (PatientsLikeMe) to assist Veterans with epilepsy. The hypothesis is that the online social media platform, PatientsLikeMe, will improve selected patient-reported outcomes on perceived self-management skills for patients who engage in the website functions.

ELIGIBILITY:
Inclusion Criteria:

* US Veteran
* Epilepsy (Seizure Disorder)
* >18 years

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Epilepsy Self-Management | 6 weeks
  The Epilepsy Self-Management Scale (ESMS) is a 38 item scale that assesses "frequency of use of epilepsy self-management practices." A 5-point Likert scale asks participants to respond from never to always. The scale includes 5 subscales that measure medication management, Information management, Safety management, Seizure management, and Lifestyle Management. Higher scores indicate more frequent use of self-management strategies. The scale and its subscale have been previously validated and used in similar studies.
Epilepsy Self-Efficacy | 6 weeks
  The Epilepsy Self-Efficacy Scale is a 33-item scale that measures "aspects of efficacy in the self-management of epilepsy". An 11-point Likert rating scale asks participants to choose from 0, I cannot do at all to 10, sure I can do. The scale contains three dimensions: 1) self-efficacy for medication management, 2) self-efficacy for seizure management and 3) self-efficacy for general management issues. Higher scores correspond to higher levels of self-efficacy. The scale has been validated and used in similar studies of website interventions for epilepsy patients.

SECONDARY OUTCOMES:
Epilepsy Self-Management Information Scale | 6 weeks
  This is a subscale of the Epilepsy Self-Management Scale, which measures the frequency with which patients use strategies to manage information about their epilepsy

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States